CLINICAL TRIAL: NCT04339114
Title: Reason to Season; Flavors to Increase Vascular Health
Acronym: SPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB 2019-014
Record Dates: First submitted 2020-04-06; First posted 2020-04-09 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Overweight and Obesity; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control meal (Sham Comparator): Pancake
  Interventions: Other: Breakfast: control meal
- Control meal + Cinnamon (Active Comparator): Pancake seasoned with cinnamon
  Interventions: Other: Breakfast: Cinnamon meal
- Control meal + Italian herb mix (Active Comparator): Pancake seasoned with Italian herb mix
  Interventions: Other: Breakfast: Italian herbs meal
- Control meal + Active-Herbs/Spice mix (Active Comparator): Pancake seasoned with pumpkin spice
  Interventions: Other: Breakfast: pumpkin spice

INTERVENTIONS:
Other: Breakfast: control meal — The breakfast meal includes a Taiwanese style pancake plus a side of hash browns with ketchup. Every meal will be individualized to meet the 30% of the energy requirement of subjects based on the Harris benedict equation.
  Arms: Control meal
Other: Breakfast: Cinnamon meal — The breakfast meal includes a Taiwanese style pancake seasoned with grounded cinnamon plus a side of hash browns with ketchup. Every meal will be individualized to meet the 30% of the energy requirement of subjects based on the Harris benedict equation.
  Arms: Control meal + Cinnamon
Other: Breakfast: Italian herbs meal — The breakfast meal includes a Taiwanese style pancake seasoned with Italian herbs plus a side of hash browns with ketchup. Every meal will be individualized to meet the 30% of the energy requirement of subjects based on the Harris benedict equation.
  Arms: Control meal + Italian herb mix
Other: Breakfast: pumpkin spice — The breakfast meal includes a Taiwanese style pancake seasoned with pumpkin spices plus a side of hash browns with ketchup. Every meal will be individualized to meet the 30% of the energy requirement of subjects based on the Harris benedict equation.
  Arms: Control meal + Active-Herbs/Spice mix

SUMMARY:
Scientific evidence is growing on the health benefits of herbs/spices. The study is interested in understanding how various herb and spice blends influence the function of blood vessels. The study is also interested in how blood sugar, the insulin hormone and immune cells may be related to how well the blood vessels function. Herbs and spices have components called phytochemicals that may be related to how well blood vessels function. The study is planned to investigate these relationships.

After qualifying to participate in the research study, participants will be asked to come to the Clinical Nutrition Research Center (CNRC) for four on-site Study Days, each lasting for about 8 hours with a 40 min followup to measure vessels' function the next morning. On each Study Day, different amounts of herbs/spices will be included in a breakfast meal. The herbs and spices are purchased in the grocery store and are Italian herbs, cinnamon, and a mix of pumpkin pie spices (cinnamon, ginger, clove, nutmeg).

All meals will be prepared in the CNRC's kitchen using foods and ingredients purchased at the local grocery store. Blood collection and blood vessel function tests will be performed during the Study Day using typical procedures used in hospitals, doctor offices, and clinics.

DETAILED DESCRIPTION:
This clinical trial is a single-center randomized, blinded, multi-arm, within subjects, cross over design and features a repeated postprandial sampling paradigm to evaluate the effects of herbs/spices on vascular function in individuals who are overweight or moderately obese after consuming a standardized challenge meal. Subjects will undergo 4 Study Days at least 3 days apart. On each Study Day subject will receive a standardized meal made with: salt and pepper only (Control condition) or the same meal with up to 6 gram herbs/spice mix or Italian herb mix or cinnamon.Each Study Day will last about 8 h with a 40 min follow up the following morning to complete a 24 h set of procedures. The 24 h assessment allows for assessment of clinical effects over an extended time frame.

STUDY PROCEDURES:

1. Screening Visit:

   Interested subjects will be asked to come to the Clinical Nutrition Research Center (CNRC) on the IIT (Illinois Tech) Campus, Chicago, IL, where the study will take place for all in person visits. The screening visit is the first visit and will be used to determine if an interested person is eligible to participate in the study. The screening visit will take 2 hours. Prospective subjects must read, sign and date a written Institutional Review Board approved Informed Consent Form prior to performing any study procedure. One of our Study investigators will go through the inform consent (ICF) with subject comprehensively to explain all study related activities as mentioned in the ICF form.

   At the on-site screening visit, subject will be asked to arrive after overnight fasting for 10-14 hours and be well-hydrated. Subjects will be instructed to drink plenty of water the 24 hours before the screening visit to ensure they are well hydrated (ie., aim for intake of at least 8-10 cups over 24 h). They will also be asked to abstain from vigorous exercise 12 h before the visit. Light activity is acceptable. A series of procedures will be conducted to determine eligibility to participate in the study, including venous or capillary blood sampling (by finger prick) to test blood glucose (to ensure fasting status and inclusion criteria), anthropometric measurements (height, weight, waist circumference, body composition), Body Mass Index (BMI, calculated from height and weight) calculation, vital sign measurements (blood pressure and heart rate), body temperature measurement (by ear thermometer), and completion of a series of questionnaires relating to their general health and lifestyle. For vital sign measurements, subjects will sit in a comfortable chair, feet uncrossed and on the floor and will be asked to rest quietly for 5 minutes before measuring blood pressure and heart rate. Arm vein will be assessed using a vein access scale test.

   Based on the results of fasting blood glucose concentration, the questionnaires, and health evaluation, subjects who meet the inclusion and none of the exclusion criteria will be invited to participate in the study.

   Subjects who are eligible and accept the invitation to participate will be counseled on following a limited polyphenolic diet throughout the duration of their participation, although more strict guidelines will be imposed during the 3 days prior to each study visit. Shopping lists and meal plans will be provided to subjects, along with counseling by our staff, to help subjects adhere to the limited polyphenolic diet. Subjects will be asked not to take any allergy medications and/or any pain medications such as Aspirin, Excedrin, Ibuprofen (Advil, Motrin, Nuprin), Naproxen, Aleve within 48 hours of each scheduled study days. Tylenol is allowed. The visit will be rescheduled when allergy/pain medication is needed within 48 hours prior to study days.

   Before leaving the CNRC, subjects will be provided instructions for "How to prepare for study day", which will include avoidance of vigorous physical activity and alcoholic beverages, and caffeinated beverages at least 24 hours preceding a Study Day. Usual coffee and tea can be consumed up to noon time the day before and water encouraged thereafter. Subjects will also be encouraged to get a usual night of sleep and maintain usual dietary patterns, except for the guidance provided for limited polyphenol foods and beverages.
2. Study Day Three days prior to each Study Day, subjects will be instructed NOT to consume berry containing foods, or dark chocolate and record 3-consecutive days of food intake. Subjects will be instructed to consume a usual dinner meal the night before the Study Day and be required to repeat the same dinner and afternoon snacks the night before the second, third and fourth Study Days.

On each Study Day, subjects will arrive at the clinic after fasting for 10-14 hours and in a well-hydrated and well-rested state. If they are taking any medication(s) on regular basis, they will be asked not to take the medication(s) at home and instead bring to the CNRC to be taken in the presence of the study investigator so the medications(s) is taken at the same time before each Study Day visit.

On the Study Day, after confirming compliance with the pre-study day procedures, anthropometric measurements, vital signs (blood pressure, heart rate and ear temperature) and capillary blood sampling (finger prick, confirmation of fasting state) will be taken. A licensed healthcare professional (LHCP) will evaluate and place an intravenous catheter at the antecubital site of subject's arm. An intravenous catheter is a thin flexible tube that allows sampling of blood through one port throughout the Study Day. Once the catheter is placed, a baseline blood sample will be taken (Time point t=0).

After completing a baseline blood draw, flow-mediated dilation (FMD) procedure will be measured. Afterwards, subjects will receive a breakfast meal along with a drink beverage (Control meal, Control meal +Active-Herbs/Spice mix, or + Italian herbs mix, or +Cinnamon). The first blood sample will be collected at 0h, with FMD and additional blood samples conducted/collected at 0.5h, 1 h, 2h, 4h, 5.5h, and 7h. After completion of the 7h blood collection and FMD procedure, the catheter will be removed and subjects will be evaluated for safety and/or discomfort/symptoms and they will be given a take-home snack. Subjects will be asked to return the next morning for completion of 24 h procedures. All dinner and afternoon snacks consumed on Study Day will be asked to be repeated for future Study Days.

Blood collection: There will be a total of 8 times of blood collection for each Study Day. At the 0h, 2h, 4h, and 7h time points, blood will be collected a total of 64 milliliters (mL) (16 mL per each time point) of blood. At the 0.5 h, 1 h, 5.5 h and 24h time points, a total of 32 mL (8 mL per each time point) of blood will be collected. The total amount of blood collection per test day 96 mL. . During the whole study, total amount of 384 mL of blood will be collected which is less than the amount allowed for one time blood donation(550mL).

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 25 and 35 kg/m2
* Aged over 18 years old
* Able to provide informed consent and comply with study procedures
* Willing to maintain stable body weight and follow his/her habitual diet and physical activity patterns throughout the trial.
* People with no documented disease condition that would interfere with the study endpoints (ie., Cardiovascular disease (CVD), diabetes, hypertension (diagnosed high blood pressure), major organ diseases) or taking medication or dietary supplements that may interfere with study endpoints.
* Judged by the Investigator to be in general good health on the basis of medical history and screening laboratory tests.
* Premenopausal women are studied at the same time of the month during the follicular phase of their menstrual cycle (first 14 days of cycle).

Exclusion Criteria:

* Current smoker and/or marijuana user, past smokers may be allowed in the study if stopped >2 years
* Have a history or presence of atherosclerotic cardiovascular disease, inflammatory disease, diabetes mellitus, or other systemic diseases, psychological or psychiatric disorders that may interfere with study outcomes
* Unstable use of any medication/supplement - Have a history of cancer, except for non-melanoma skin cancer within past 5 years
* Addicted to drugs and/or alcohol (>4 drinks/day)
* Have been exposed to any non-registered drug product within last 30 days.
* Working overnight (e.g. 3rd shift of overnight workers)
* Have allergies/intolerances to cinnamon, Italian herbs, or other spices or study foods
* Excessive exercisers or trained athletes
* Extreme dietary habits (i.e., vegan)
* Excessive coffee/tea drinker (> 4cups/day)
* Actively losing weight/ trying to lose weight (unstable body weight fluctuations of > 5 kg in 3 months)
* Donated blood within last 3 months
* Female who is pregnant, planning to be pregnant, or breastfeeding
* The individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
To characterize the time course of herbs/spice action on endothelial function as measured by Flow Mediated Vasodilation (FMD) over 24 h using a challenge meal paradigm individualized per subject energy requirements to maintain body weight. | Baseline(T0)-24 hours
  Flow mediated vasodilation (FMD): Ultrasound imaging of the brachial artery is a non-invasive technique that assesses endothelial-dependent relaxation and is used as a surrogate marker of large vessel (macrovascular) endothelial function. FMD will be studied in the brachial (arm) artery of all subjects using standardized methods recommended by the American College of Cardiology

SECONDARY OUTCOMES:
Changes in plasma glucose concentration-response between 4 treatments | Baseline(T0)-24 hours
  Plasma glucose concentration will be measured using Randox Daytona automated Clinical Analyzer.
Changes in plasma insulin concentration-response between 4 treatments | Baseline(T0)-24 hours
  Plasma insulin concentration will be measured using Randox Daytona
Changes in inflammation signaling response between 4 treatments | Baseline (T0)-7 hours
  Peripheral Blood mononuclear cells will be tested using immunocytochemistry.

OTHER OUTCOMES:
To assess effects of herbs/spices on inflammatory markers | Baseline (T0)-24 hours
  Plasma cytokines IL-6 concentration will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Insititute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States